CLINICAL TRIAL: NCT07356349
Title: AuthenTicity of Point of Care Urine samplEs Using Oral fluoreScein Sodium in adulTs With substancE Use Disorder
Brief Title: Study to Confirm the AuthenTicity of Point of Care Urine samplEs Using Oral fluoreScein Sodium in adulTs With substancE Use Disorder (ATTESTED)
Acronym: ATTESTED
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UpTru Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: UPTRu-301
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorder (SUD)
Keywords: randomized controlled trial; substitution heuristic
MeSH Terms: conditions — Substance-Related Disorders | interventions — Fluorescein

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluorescein (Experimental): Ingestion of 100 mg of fluorescein with 250 ml Gatorade tm
  Interventions: Drug: Fluorescein
- placebo (Placebo Comparator): ingestion of 250 ml Gatorade tm without fluorescein
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Fluorescein — Oral ingestion of 100 mg of fluorescein in 250 ml of Gatorade tm
  Other Names: Experimental: Fluorescein
  Arms: Fluorescein
Other: placebo — Ingestion of 250 ml of Gatorade tm without fluorescein
  Arms: placebo

SUMMARY:
The purpose of this phase III, randomized, double-blind, placebo-controlled study is to confirm the authenticity of point-of-care urine samples in adult persons with substance use disorder using fluorescein sodium as a marker. Eligible persons will, drink a sample of Gatorade™ which includes either, 100 mg fluorescein sodium, or not, followed by 500 mL of water. Fifteen minutes after consuming the Gatorade™, participants will provide a mid-stream urine sample (at least 10 mL urine is required) for examination of fluorescence (in a single-blinded manner) using a Qubit™ fluorometer.

DETAILED DESCRIPTION:
One hundred fourteen eligible persons will be randomized. One hour after completely emptying their bladders, in a blinded manner, half will receive Gatorade and the other half will receive Gatorade with 100 mg of fluorescein. All will then drink 500 ml of water and 15 minutes later they will provide urine samples. A solution of sodium bicarbonate will be added to the samples and blinded observers will then examine all of the samples for fluorescence using a Qbit fluorometer.

ELIGIBILITY:
Inclusion Criteria:

* • Written informed consent, obtained from the person or legally acceptable representative, before any study-related procedure is performed. Adults aged between 18 and 65 years, inclusive, at the time of signing the informed consent form.

  * A documented current substance use disorder, including but not limited to alcohol, cocaine, and/or opioid.
  * Female participants must be: Not women of childbearing potential (WOCBP), i.e., postmenopausal and/or surgically sterile, OR: WOCBP who agree to use a contraceptive method that is highly effective (based on the investigator's judgment) for 28 days before and after study product administration.
  * Male participants must agree to use effective birth control methods and must not donate sperm until 2 weeks after study product administration.
  * Must agree not to be a gamete donor from Screening until 28 days after the follow-up telephone call.
  * Willing and able to comply with the study instructions and attend all scheduled study visits.

Exclusion Criteria:

* Life expectancy less than 5 years.

  * Women who are pregnant or are breast-feeding.
  * Known cirrhosis.
  * Diagnosis of Gilbert's syndrome.
  * Heart failure, classified as being in New York Heart Association Class II-IV at Screening.
  * Known allergy to fluorescein, Gatorade™, or any of their excipients.
  * Estimated glomerular filtration rate <30 mL/min/1.73m2 using the Cockroft-Gault method at Screening.
  * Hemoglobin <120 g/L at Screening.
  * Diagnosis of sickle cell anemia or sickle cell trait.
  * Any major episode of infection requiring hospitalization and/or treatment with intravenous antiinfective agents during the 2 months prior to Screening.
  * Use of fluorescein for medical imaging (eg, angiogram, corneal staining) in the 3 days prior to the Randomization Visit. UP
  * In the opinion of the investigator, any other condition that would preclude participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection | 15 minutes post ingestion
  Presence of fluorescence
Detection | 15 minutes post ingestion
  Presence of fluorescence .30,000 using fluorometer

IPD SHARING:
Plan to Share IPD: Yes
raw data & analysis-ready data sets
Time Frame: start date :January 1 2028 end date : December 31 2030
Access Criteria: Researchers who confirm that the data will be only used for medical scientific purposes, as per World Medical Association Helsinki Declaration 2024 will be able to submit their coordinates, and the data sets will be shared with them.
URL: https://www.uptru.com

REFERENCES:
- See also: Sponsor's Home Page — https://www.uptru.com/
- See also: Related Info — https://www.uptru.com/